CLINICAL TRIAL: NCT06957106
Title: Myocardial Injury in Geriatric Patients Followed in Intensive Care Unit After Noncardiac Surgery
Brief Title: Myocardial Injury Noncardiac Surgery in Geriatric Patients
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Berkehan Nizamlıoğlu, resident doctor, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: FSMTRH-MBN-02
Record Dates: First submitted 2025-04-21; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-01

CONDITIONS: Myocardial Injury After Noncardiac Surgery (MINS)
Keywords: myocardial injury; intensive care unit; geriatric patients; troponin elevation; ICU outcomes; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric ICU Patients: Geriatric patients (aged ≥65 years) who underwent surgery under general or regional anesthesia and were admitted to the intensive care unit in the postoperative period between January 2018 and August 2023.

SUMMARY:
In inpatients aged 45 years and older, the approximate peri-operative mortality rate after non-cardiac surgery is around 1% to 2%. Half of these deaths are attributed to cardiovascular complications of surgery. Postoperative cardiac troponin elevation with ≥1 measurement of cardiac troponin ≥99% percentile above the upper limit of the reference value, which is an indicator of acute myocardial injury, is seen in the first 30 days after surgery and usually occurs within 72 hours. Myocardial damage is thought to result from an ischemic mechanism. Clinical symptoms may be masked by sedation or analgesia in the perioperative period, so evidence of an ischemic feature (e.g. ischemic symptoms, electrocardiographic changes) is not required. These criteria are defined as MINS (Myocardial Injury Non Cardiac Surgery) criteria. In this study, the investigators aimed to investigate the intensive care follow-up processes and outcomes of geriatric patients over 65 years of age in whom MINS was detected during postoperative intensive care monitoring.

DETAILED DESCRIPTION:
In this study study, 117 geriatric patients aged ≥65 years who were followed and treated in the intensive care unit in the postoperative period after general or regional anesthesia between January 2018 and August 2023 after obtaining Ethics Committee Approval (FSM EAH-KAEK 2023/140) were retrospectively analyzed. Age, gender, comorbidities, coronary artery disease, heart failure, atrial fibrillation, history of chronic renal failure, presence of emergency surgery, preoperative antiaggregant use, ASA score, type of surgery, presence of laparoscopic or open surgery, anesthesia and duration of surgery, intra operatively; hypotension, tachycardia, bradycardia, presence of blood and blood products transfusion, duration if hypotension developed, first day of intensive care unit hospitalization; APACHE, SAPS, SOFA scores, duration of mechanical ventilation, presence and duration of troponin elevation, the day of hospitalization, if cardiac examination was performed; Ejection fraction, diastolic dysfunction, presence of revascularization treatment, hemoglobin, hematocrit levels on the day of troponin elevation, neutrophil/lymphocyte ratio, procalcitonin, crp levels, use of antiaggregants, mechanical thrombophylaxis, acidosis, presence of hypoxia, need for vasopressor therapy, type of discharge from intensive care unit and presence of mortality will be recorded

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or older
* Patients who underwent major, moderate, or minor surgery under general and/or regional anesthesia
* Patients who were followed and treated in the postoperative intensive care unit

Exclusion Criteria:

* Patients younger than 65 years of age
* Patients with preoperative troponin levels above the normal reference range
* Patients with active myocardial ischemia symptoms (e.g., chest pain, pain radiating to the neck, jaw, shoulder, or arm)
* Patients with known pre-existing cardiac disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study includes geriatric patients aged 65 years and older who underwent major, moderate, or minor surgery under general and/or regional anesthesia and were followed postoperatively in the intensive care unit between January 2018 and August 2023 at Fatih Sultan Mehmet Training and Research Hospital. The study population consists of patients whose medical records were retrospectively reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
30-day postoperative mortality | 30 days
  Association between postoperative troponin elevation and ICU mortality in geriatric patients. Mortality status recorded in hospital database

SECONDARY OUTCOMES:
mechanical ventilation | 30 days
  Duration of mechanical ventilation in patients over 65 years of age with postoperative mins.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Yildirim Ar, As Prof, Study Director — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital,, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This is a retrospective observational study. Individual participant data will not be shared.

REFERENCES:
- [Background] Gao L, Chen L, He J, Wang B, Liu C, Wang R, Fan L, Cheng R. Perioperative Myocardial Injury/Infarction After Non-cardiac Surgery in Elderly Patients. Front Cardiovasc Med. 2022 May 19;9:910879. doi: 10.3389/fcvm.2022.910879. eCollection 2022. PMID 35665266
- [Background] Park J, Lee JH. Myocardial injury in noncardiac surgery. Korean J Anesthesiol. 2022 Feb;75(1):4-11. doi: 10.4097/kja.21372. Epub 2021 Oct 18. PMID 34657407
- [Background] Ruetzler K, Smilowitz NR, Berger JS, Devereaux PJ, Maron BA, Newby LK, de Jesus Perez V, Sessler DI, Wijeysundera DN. Diagnosis and Management of Patients With Myocardial Injury After Noncardiac Surgery: A Scientific Statement From the American Heart Association. Circulation. 2021 Nov 9;144(19):e287-e305. doi: 10.1161/CIR.0000000000001024. Epub 2021 Oct 4. PMID 34601955